CLINICAL TRIAL: NCT05903950
Title: Air Pollution and Cardiovascular Disease in Qatar: an Interventional Study to Reduce Blood Pressure: the APCIQ-BP Trial
Brief Title: Air Pollution and Cardiovascular Disease in Qatar: an Interventional Study to Reduce Blood Pressure
Acronym: APCIQ-BP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Cornell Medical College in Qatar (Other)
Collaborators: Hamad Medical Corporation (Industry); Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 22-00009
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Hypertension, Systolic; Metabolic Syndrome
Keywords: hypertension; metabolic syndrome; air pollution
MeSH Terms: conditions — Isolated Systolic Hypertension; Metabolic Syndrome; Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active mode (Active Comparator): In home use of portable air cleaners with a High Efficiency Particulate Air (HEPA) filter for 4 weeks.
  Interventions: Device: Air cleaners with HEPA filter
- Sham mode (Sham Comparator): In home use of portable air cleaners without a High Efficiency Particulate Air (HEPA) filter for 4 weeks.
  Interventions: Device: Air cleaners without HEPA filter

INTERVENTIONS:
Device: Air cleaners with HEPA filter — PM 2.5 exposure reduction using in home portable air cleaners fitted with HEPA filters
  Arms: Active mode
Device: Air cleaners without HEPA filter — Simulation of PM 2.5 exposure reduction using in home portable air cleaners without HEPA filters.
  Arms: Sham mode

SUMMARY:
The main objective is to determine if in-home portable air cleaners provide persistent reductions in PM2.5 exposures and improvements in systolic blood pressure and biochemical parameters over 4-weeks in patients with metabolic syndrome residing in Qatar.

DETAILED DESCRIPTION:
Chronic cardio-metabolic diseases such as hypertension and diabetes contribute disproportionately to global morbidity and mortality and are increasing believed to have multiple environmental influences.

PM2.5 is the fifth leading risk factor for global mortality - largely due to cardiovascular disease (CVD). Reducing personal exposure to air pollution has shown promise in improving key cardiovascular risk factors (blood pressure and insulin resistance) in limited studies, but durability of these effects is not known. Personal air cleaners have been shown to decrease personal exposure to PM2.5 and reduce blood pressure in small studies and may serve as a pragmatic intervention in high-risk patients in whom air pollution is a strong contributor to cardiovascular health.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers (100% abstinence from use of any smoking or vaping product during the prior year)
* Age ≥18 and less than 60 years old
* Living in a single residence (home, apartment) located anywhere in Qatar
* Mild systolic hypertension: screening visit systolic BP 130 to 159 mm Hg (off treatment or taking ≤ 2 BP medications that have been stable without changes during prior 4 weeks) plus ≥ 2 more additional criteria for the metabolic syndrome:

  * Waist circumference ≥102 cm if male and ≥88 cm if female
  * Fasting triglycerides ≥150 mg/dL (or taking a triglyceride-lowering medication)
  * HDL-C ≤ 40 mg/dL if male and ≤ 50 mg/dL if female (or taking an HDL-raising medication),
  * Fasting glucose ≥100 mg/dL

Exclusion Criteria:

* Pregnancy (self-reported)
* Screening visit urine positive for cotinine (NicAlert >100 ng/mL)
* Living with an active smoker who smokes indoors (by self-report)
* High risk conditions that prohibit allowing home BP to be >130/80 mm Hg during the10-week trial including any cardiovascular disease (coronary artery disease, prior stroke, heart failure, peripheral arterial disease, aneurysm) or ≥ stage 3 kidney disease (estimated glomerular filtration rate < 60 ml/min)
* A medical condition placing the participant at risk from participation (per investigators)
* Expected overnight travel outside their residence during the study
* HEPA filter within the air conditioners of the residence (self-reported) or individual use of HEPA filter
* Unable to comprehend/sign an informed consent
* Lung disease requiring oxygen
* Cancer receiving treatment
* Screening visit: BP ≥160/100 mm Hg or fasting blood glucose ≥126 mg/dL and confirmed diabetes with follow-up HbA1c ≥6.5%. If glucose is elevated ≥126 mg/dL but HbA1c<6.5%, they could still participate.
* Medication changes in past 4 weeks. If participants are on medications for high BP or hyperlipidemia, they will need to have had stable therapy during prior 10 weeks with no planned changes during the study
* Left upper arm circumference >17 inches as this will make BP levels inaccurate with the home monitor used
* Acute illness or infectious symptoms within the prior 4 weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-03 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure | week 4, week 10
  Mean change from baseline in systolic blood pressure

SECONDARY OUTCOMES:
Change in Fasting Glycemia | week 4, week 10
  Mean change from baseline in fasting glycemia
Change in Insulin Resistance Index | week 4, week 10
  Mean change from baseline in Insulin Resistance Index

CONTACTS AND LOCATIONS:
Overall Officials: Charbel Abi Khalil, MD, Principal Investigator — Weill Cornell Medical College in Qatar
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after de-identification (test, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately after publication. No end date.
Access Criteria: Anyone who wishes to access the data